CLINICAL TRIAL: NCT00013351
Title: Restricted Useful Field View as a Risk Factor in Older Adults
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: C1830R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Vision Impairment
Keywords: Aging adult, attention, falls, vision
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Prevention of Falls

SUMMARY:
The relationship between Useful Field of Vision (UFOV) and falls taken by the elderly will be investigated. UFOV is a test which measures visual attention. The test has been used in correlating the visual attention in the elderly with their driving safety record. The test is administered using a computer and consists of three parts: a) subject views figures which appear in the center of the computer screen and identified them as quickly as possible; b)the subject has to identify figures in the center of the screen while at the same time point to another symbol which will appear in one of eight places on the outer portion of the screen; c) the third section is similar to the second except while the subject is identifying and pointing there is a background noise.

ELIGIBILITY:
Vision impaired adults at risk for falls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1998-04; Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Decatur, Decatur, Georgia, United States